CLINICAL TRIAL: NCT02120053
Title: Interest of Bone Substitute Material in Immediate Complete Denture: a Controlled Randomized Clinical Trial
Brief Title: Interest of Bone Substitute Material in Immediate Complete Denture
Acronym: PANORAMIX
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P111116; AOR12032 (Other: APHP sponsor)
Record Dates: First submitted 2014-04-15; First posted 2014-04-22 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Alveolar Bone Loss; Denture Complete Immediate; Bone Substitute; Replacement Material; Bone
Keywords: Immediate complete denture; Alveolar ridge resorption; Alveolar bone loss; Bone substitute material; Edentulism
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone substitute material group (Experimental): Immediate denture placement following extractions and alveolar sockets filling with bone substitute material
  Interventions: Device: Bone substitute material group
- Conventional protocol (Active Comparator): Immediate denture placement following the conventional protocol
  Interventions: Device: Conventional protocol

INTERVENTIONS:
Device: Conventional protocol — Teeth extractions and conventional immediate complete denture placement
  Arms: Conventional protocol
Device: Bone substitute material group — Teeth extractions and sockets filling with bone replacement material before immediate complete denture placement
  Arms: Bone substitute material group

SUMMARY:
More than 2 million French people suffer from the widespread disability of edentulism, with large consequences on function, nutrition, aesthetics and well-being. Complete denture is a common therapeutic strategy.

The immediate complete denture technique consists in placing the denture in the same clinical session as last anterior teeth extractions. With this technique, aesthetic and function are immediately reintroduced and the patient is never left toothless or without any denture.

After teeth extractions, alveolar healing process leads to ridge resorption with bone volume modifications and reduction in height and width.

However ridge bone volume is an essential factor in removable denture stability. With implantology as an alternative prosthetic strategy, ridge volume is also a most important factor to place dental implants in a situation close to previous dental roots position. In order to preserve bone volume, a current alternative strategy proposes to place bone substitute materials in tooth sockets after extraction. This strategy was never evaluated with the immediate complete denture technique.

Hypothesis: A new strategy associating immediate complete denture and bone substitute material is more effective than conventional immediate complete denture in a bone preservation perspective.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for maxillary immediate complete denture, presenting a Kennedy
* Class I partial dentition (bilateral posterior tooth loss)
* Over 18 years of age
* Healthy adhering gingiva
* Willing to participate in the study, able to sign the consent form

Exclusion Criteria:

- Medical conditions contraindicating oral surgery: progressive cancer history of radiotherapy in the head and neck region major neurological disease anti-coagulant treatment with prothrombin time<30% valvulopathy, hematologic disease, agranulocytosis, serious heart failure, recent myocardial infarction < 5 years immune deficiency, AIDES osteomalacia hepatic or renal insufficiency unregulated diabetes long-term steroids treatment bisphosphonates

* Allergy to collagen
* Pregnant or nursing women
* Persons specially protected
* Non-affiliated with the social security system persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of bone ridge height one year after maxillary immediate complete denture placement with or without bone substitute material in incisive-canine sockets | one year (365 days)

SECONDARY OUTCOMES:
Height and width average between day 10th and day 90th after maxillary immediate complete denture placement, and between day 10th and one year | Day 10, Day 90, Day 365
  To compare bone ridge width one year after maxillary immediate complete denture placement with and without bone substitute material in incisive-canine sockets: height and width average between day 10th and day 90th after maxillary immediate complete denture placement, and between day 10th and one year

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Rignon-Bret, DDS, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Background] Tallgren A, Lang BR, Walker GF, Ash MM Jr. Roentgen cephalometric analysis of ridge resorption and changes in jaw and occlusal relationships in immediate complete denture wearers. J Oral Rehabil. 1980 Jan;7(1):77-94. doi: 10.1111/j.1365-2842.1980.tb01466.x. PMID 6987348
- [Background] Park JB. Healing of extraction socket grafted with deproteinized bovine bone and acellular dermal matrix: histomorphometric evaluation. Implant Dent. 2010 Aug;19(4):307-13. doi: 10.1097/ID.0b013e3181e5abbc. PMID 20683287
- [Background] Araujo MG, Liljenberg B, Lindhe J. Dynamics of Bio-Oss Collagen incorporation in fresh extraction wounds: an experimental study in the dog. Clin Oral Implants Res. 2010 Jan;21(1):55-64. doi: 10.1111/j.1600-0501.2009.01854.x. PMID 20070748
- [Background] Rignon-Bret C, Rignon-Bret JM. Prothèse amovible complète, prothèse immédiate, prothèse supra-radiculaire et implantaire. Ed CdP, Collection JPIO 2002.
- [Derived] Rignon-Bret C, Hadida A, Aidan A, Nguyen TH, Pasquet G, Fron-Chabouis H, Wulfman C. Efficacy of bone substitute material in preserving volume when placing a maxillary immediate complete denture: study protocol for the PANORAMIX randomized controlled trial. Trials. 2016 May 20;17(1):255. doi: 10.1186/s13063-016-1380-7. PMID 27206923